CLINICAL TRIAL: NCT04607824
Title: Computational Task in Duchenne Muscular Dystrophy: Involvement of Cardiac Autonomic Regulation.
Brief Title: Heart Rate Variability in Duchenne Muscular Dystrophy During Computer Task
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carlos Bandeira de Mello Monteiro, Associate Professor, University of Sao Paulo
Other Study IDs: 14508213.4.0000.0065
Record Dates: First submitted 2020-10-22; First posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Heart rate variability; Duchenne muscular dystrophy; Typically developed; Autonomic nervous system; Chaotic global techniques
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Duchenne Muscular Dystrophy group: Forty-five male subjects were included in the Duchenne Muscular Dystrophy (DMD) group and they were assessed for twenty minutes at rest sitting, and then five minutes whilst performing the maze task on a computer.
  Interventions: Behavioral: Duchenne Muscular Dystrophy group
- Typical Development group: Forty-five male subjects were included in the healthy Typical Development (TD) control group and they were assessed for twenty minutes at rest sitting, and then five minutes whilst performing the maze task on a computer
  Interventions: Behavioral: Typical Development group

INTERVENTIONS:
Behavioral: Duchenne Muscular Dystrophy group — Assessment of heart rate variability at rest and during computational task in people with Duchenne muscular dystrophy
  Groups: Duchenne Muscular Dystrophy group
Behavioral: Typical Development group — Assessment of heart rate variability at rest and during computational task in people with typical Development
  Groups: Typical Development group

SUMMARY:
HRV is attained using a Polar RS800CX. Then, evaluated through linear, non-linear and chaotic global techniques (CGT). Forty-five male subjects were included in the DMD group and age-matched with forty-five in the healthy Typical Development (TD) control group. They were assessed for twenty minutes at rest sitting, and then five minutes whilst performing the maze task on a computer.

DETAILED DESCRIPTION:
This is a cross-sectional study, where HR was recorded beat-to-beat (RR intervals) using the portable Polar RS800CX HR monitor (Polar Electro, Finland). HR was recorded before the onset and at the end of the five minutes of the computer maze paradigm task.

The subjects were seated in a standard chair (walkers, TD group and DMD) or in their own wheelchair (non-walkers, DMD group), the Polar watch was positioned on the wrist. The analysis of HRV was possible through the recording of RR interval in two periods: the period of twenty minutes at seated rest, and then during the computer task for five minutes.

The computer task used a maze paradigm with one correct pathway that could be negotiated and ultimately solved. All participants were positioned comfortably and an evaluator responsible for instruction and annotation of data.

Each individual was instructed to walk the correct path with the digital character pawn (pointed on the screen by the evaluator) to the exit of the maze identified by an "x" (pointed on the screen by the evaluator). It was provided for the subjects, who used the arrow buttons on the keyboard, identified by up, down, right and left, using the dominant hand, with the arrows moving through a 20 x 20 cm maze. Participants were requested to complete the maze as fast as possible.

HRV analysis followed the guidelines published by the Task Force of the European Society of Cardiology and North American Society of Pacing and Electrophysiology. The RR intervals were recorded, and then were downloaded to the Polar Precision Performance program (v.3.0). This software enabled the visualization of HR and the extraction of a cardiac period (RR intervals series; the variation of beat-to-beat interval in milliseconds) file in ".txt" format. For analysis of HRV data at rest, we analyzed 1000 consecutive RR intervals, and for HRV analysis for the computational task, the number of consecutive RR intervals obtained was exactly 256 RR intervals. Digital filtering complemented by manual filtering was performed to eliminate artifacts and only series with greater than 95% of sinus beats were included in the study. HRV analysis was undertaken through linear, non-linear and chaotic global techniques (CGT).

ELIGIBILITY:
Inclusion Criteria:

* DMD diagnoses was based on molecular methods and/or muscular protein expression.
* TD age-matched with DMD.

Exclusion Criteria:

* subjects with severely dilated myocardium.
* subjects with other associated diseases.
* individuals with inability to understand task instructions.

Ages: 9 Years to 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 45 individuals with DMD (convenience sample) and 45 age-matched healthy TD individuals participated in the trial.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability behavior during computational task | 1 day
  Linear, non-linear and complexity indices of heart rate variability will be assessed at rest and during computational task, in order to analyse it's behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos BM Monteiro, Ph.D., Principal Investigator — University of Sao Paulo
Locations (1):
- Comitê de ética da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided